CLINICAL TRIAL: NCT04704583
Title: Parental Guidance for Parents of Highly Dependent Adult Children
Brief Title: Parental Guidance for Failure to Launch.
Acronym: SPACE-FTL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000029082; No NIH funding (Other: 01.18.24)
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Failure to Launch; Anxiety Disorders; Hikikomori
Keywords: Parents; Child
MeSH Terms: conditions — Anxiety Disorders; hikikomori

STUDY DESIGN:
Intervention Model Description: randomized wait-list control group design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (active) (Experimental): Individuals in this group will start treatment after the initial assessment, without a delay.
  Interventions: Behavioral: SPACE parental-guidance
- Wait-list control group (Active Comparator): Individuals in this group will start treatment after the initial assessment, with a delay of thirteen weeks.
  Interventions: Behavioral: SPACE parental-guidance

INTERVENTIONS:
Behavioral: SPACE parental-guidance — The treatment will be delivered to the parents in ten 50-minute sessions. The sessions are planned to be weekly and will be completed within 13 weeks of the first session. The sessions include instruction and education, acquiring skills, role-play, and simulations. Parents will be given exercises and goals in reducing accommodation to achieve at home (in cognitive behavioral therapy this is sometimes called 'homework') in some of the sessions. For example, parents to write down one or two things that they would most like to see their child handling better.

SUMMARY:
In the proposed study the outcome of administering parental guidance, based on the Supportive Parenting for Anxious Childhood Emotions (SPACE) program, to parents of highly dependent adult children will be explored. The proposed study's primary purpose is to assess the outcome of parental guidance. In addition, the study will also examine participants' acceptance and adherence to this parental guidance method.

DETAILED DESCRIPTION:
Recent years have seen an increase in the number of adult Americans who live with their parents. In the 18 to 34 age group, living with one's parents is currently the most common living arrangement. Some adult children have been using their parents' homes as only a temporary solution due to economic hardship. However, other adults remain at home, highly reliant on their parents, and not in higher education or employment. The latter group (who are at times referred to as 'failure to launch') are considered to suffer from a combination of a personal and familial problem and pose a significant challenge for therapists (Lebowitz, 2016). To date, little evidence exists to guide case conceptualization or intervention strategies. In this protocol, the term "FTL" for the sake of brevity in place of "highly dependent adult children who are not functioning independently" will be used.

For the clinician, work with individuals with FTL cases can seem more like treatment with child patients than adult patients. Parents often initiate clinical contact, and in many cases, the dependent adult is not open or willing to engage in treatment directly.

Dr. Lebowitz and colleagues' work with the parents of youth who suffer from clinical anxiety has suggested a theoretical conceptualization and a means of intervention in cases of FTL. Youth with anxiety display a similar pattern of reliance on parents for help in avoiding the situations they find distressing, a process known as family accommodation. Working with parents on decreasing family accommodation has been found to be efficacious in reducing anxiety and increasing independent coping in youth. This manualized approach, known as SPACE (Supportive Parenting for Anxious Childhood Emotions), has been repeatedly tested in clinical trials, including in randomized controlled trial research.

In the proposed study, the investigators will examine outcomes of a parental guidance program, based on SPACE, for parents of FTL adults (henceforth, SPACE-FTL). The current proposal builds on a published feasibility study that found reducing family accommodation was successful in FTL, and in a considerable proportion of cases the adult children started working or studying or moved to independent lodgings.

In the study, the investigators aim to investigate the SPACE-FTL outcomes including improvement in adult child symptoms and reductions in related impairment (e.g., cost-of-illness), when compared to no treatment (i.e., wait-list control). The primary hypothesis is that SPACE-FTL will decrease FTL severity and impairment, compared with the wait-list control condition. Additional outcomes will relate to the feasibility, acceptability, and parents' satisfaction of SPACE-FTL. The investigators hypothesize that parents will rate SPACE-FTL as highly acceptable and that adherence will be above 70%.

ELIGIBILITY:
Inclusion Criteria:

Individuals with FTL will be characterized as:

1. Living at parents' home.
2. Not employed gainfully for more than 10 hours per week 3. Not actively engaged in educational programs.
3. These conditions have been met for at least six months.

Participating Parents will:

1. Consent to the study and all study procedures.
2. Be proficient or fluent in English.
3. Be living with the supported individual.

Participants will be excluded based on the following conditions:

1. The individual with FTL is suffering (or likely is suffering) from a major mental disorder, per parent report. This includes any lifetime history of a psychotic disorder, bipolar disorder, Autism spectrum disorder, or intellectual delay.
2. the individual with FTL is suffering (or likely is suffering) from Substance Use Disorder (including behavioral addictions).
3. the individual with FTL has suffered a major injury or disease and thus cannot work or study.
4. The individual with FTL shows signs of acute suicidality, requiring higher level of care

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in FTL status | Once before and once after the 13 weeks of therapy
  Change in the adult child's status of accommodation, employment, and participation in academic programs. The status will be measured with the Failure to launch parent screening survey (FTL-SPS).
  FTL parent screening survey (FTL-PSS). The set of 16 screening questions builds on previous work (Hicks, 2017; Huttner, 2019; Koyama et al., 2010; Nonaka, Shimada, & Sakai, 2018; Teo et al., 2015). The questions are answered by parents/caretakers and focus on objective demographic measures of failure to launch. Parents endorse FTL-PSS items that describe their child's present FTL status.
Change in FTL symptoms | Once before and once after the 13 weeks of therapy
  Change in the adult child's status of accommodation, employment, and participation in academic programs. Symptoms will be measured with the adaptive behavior scale for Hikikomori (ABS-H).
  The Adaptive Behaviors Scale for Hikikomori (ABS-H; Nonaka et al., 2018), is a 38-item scale that measures adaptive behaviors in individuals with FTL. The scale is completed by parents. Parents answer the prevalence of symptoms on a 4 point scale (never, occasionally, often, always). A high average score indicates more FTL symptoms.
Change in clinical severity | Once before and once after the 13 weeks of therapy
  We will assess clinical severity and change in severity with the Clinical Global Impression Scale Improvement and Severity (CGI-S, CGI-I).
  Clinical Global Impression Scale - Severity (CGI-S) and Improvement (CGI-I) (NIMH, 1985). The 14-item scales will be used to assess overall severity (CGI-S) and improvement (CGI-I) at follow up visits. CGI-I scores of 1 ("very much improved") or 2 ("much improved") indicate a positive treatment response; all other responses are considered negative responses.

SECONDARY OUTCOMES:
Change in family accommodation | Once before and once after the 13 weeks of therapy
  We will measure parental accommodation with the Family Accommodation Scale - Parent Version (FASA-P)
  Family Accommodation Scale (FASA-P) (Lebowitz et al., 2013) is a self-report questionnaire used to measure accommodation of or involvement by the family in a child's anxiety symptoms. The FASA contains 9 items that rate the frequency of accommodation, the participation of parents in anxiety symptoms and changes that parents make in routines and schedules due to child's anxiety. Together these items generate the total accommodation score. One additional item assesses the degree of distress the accommodation causes the parents, and four additional items assess short-term, negative consequences of not accommodating.
Change in cost of illness | Once before and once after the 13 weeks of therapy
  We will examine changes in cost of FTL (for the individual's parents) with the Failure to Launch Cost of Illness (FTL-COI) measure.
  Cost-of-illness assessment (FTL-COI) is an in-house 14-item questionnaire that estimates the overall cost of the parent due to supporting their child. Items are summed to produce a total cost of illness per month.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data for primary and secondary measures will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available six months after study completion
Access Criteria: Data access requests will be reviewed by review panel and requestors will sign a Data Access Agreement

REFERENCES:
- [Background] Lebowitz ER, Shimshoni Y. The SPACE program, a parent-based treatment for childhood and adolescent OCD: The case of Jasmine. Bull Menninger Clin. 2018 Fall;82(4):266-287. doi: 10.1521/bumc.2018.82.4.266. PMID 30589579
- [Background] Fry, R. (2016). For First Time in Modern Era, Living with Parents Edges out Other Living Arrangements for 18-to 34-Year-Olds: Share Living with Spouse or Partner Continues to Fall. Pew Research Center.
- [Background] Lebowitz, E. R., Omer, H., Hermes, H., & Scahill, L. (2014). Parent training for childhood anxiety disorders: the SPACE program. Cognitive and Behavioral Practice, 21(4), 456-469.
- [Background] Lebowitz E, Dolberger D, Nortov E, Omer H. Parent training in nonviolent resistance for adult entitled dependence. Fam Process. 2012 Mar;51(1):90-106. doi: 10.1111/j.1545-5300.2012.01382.x. PMID 22428713
- [Background] Lebowitz ER, Woolston J, Bar-Haim Y, Calvocoressi L, Dauser C, Warnick E, Scahill L, Chakir AR, Shechner T, Hermes H, Vitulano LA, King RA, Leckman JF. Family accommodation in pediatric anxiety disorders. Depress Anxiety. 2013 Jan;30(1):47-54. doi: 10.1002/da.21998. Epub 2012 Sep 10. PMID 22965863
- [Background] Thompson-Hollands J, Kerns CE, Pincus DB, Comer JS. Parental accommodation of child anxiety and related symptoms: range, impact, and correlates. J Anxiety Disord. 2014 Dec;28(8):765-73. doi: 10.1016/j.janxdis.2014.09.007. Epub 2014 Sep 16. PMID 25261837